CLINICAL TRIAL: NCT05241548
Title: Bone Marrow Aspirate Concentrate(BMAC) on 3D Printed Polycaprolactone (PCL) Scaffold for Ridge Augmentation of Horizontal Alveolar Defects in Aesthetic Zone (Clinical Case Series Study)
Brief Title: BMAC on PCL Scaffold for Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Aly Hassan Fouad, Resident doctor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMAC 3D PCL
Record Dates: First submitted 2022-01-15; First posted 2022-02-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Bone Loss in Jaw; Edentulous Alveolar Ridge
Keywords: Ridge augmentation, BMAC , PCL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Ridge augmentation of horizontally deficient alveolar ridge in aesthetic zone by BMAC on PCL scaffold
  Interventions: Procedure: BMAC on PCL Scaffold

INTERVENTIONS:
Procedure: BMAC on PCL Scaffold — Horizontal ridge augmentation in aesthetic zone by using bone marrow aspirate concentrate on PCL scaffold

SUMMARY:
BMAC is used on 3D printed PCL scaffold for horizontal ridge augmentation in aesthetic zone , BMAC contains MSCs which can differentiate in osteogenic medium into osteoblasts which can lay down bone

DETAILED DESCRIPTION:
Alveolar bone defects were classified according to their morphology and pattern of bone loss into Class I where buccolingual loss occurs while maintaining the vertical height( Horizontal defect), Class II where vertical bone loss occurs with no buccolingual width loss (Vertical defect) and Class III where combination of vertical and horizontal bone loss occurs . These defects require augmentation before implant placement, several techniques were approached including autogenous and non autogenous bone grafting , Guided bone regeneration (GBR), ridge splitting and distraction osteogenesis. Bone grafts used with these techniques are categorized into : autografts, allografts , xenografts and alloplasts.

Autogenous bone is considered to be the gold standard in grafting because it is osteogenic in nature, osteoinductive , osteoconductive and immunologically safe The autogenous bone can be harvested intraorally from the chin area, mandibular ramus, retromolar area, maxillary tuberosity, Coronoid process, zygomatic bone or palatal and mandibular tori if present . Intraoral harvesting has the advantage of good access and no need for hospitalization but the main disadvantage is the donor site morbidity and the small amount of harvested bone. Extraoral harvesting sites include the ilium, calvarium, ribs, tibia and fibula. Extraoral harvesting solved the problem of the limited amount of harvested bone graft but the main disadvantages are the need of hospitalization, performing the harvesting procedure under general anesthesia and high morbidity due to the second surgical site Recently, tissue engineering has been used for bone regeneration so called bone tissue engineering (BTE) which aims to combine the progenitor cells to differentiate into osteoblasts, growth factors needed for regenerative process and osteoconductive scaffolds for therapeutic applications. BTE involves harvesting osteogenic cells from an autologous harvesting site ( bone marrow or adipose tissue) and/or ex vivo amplification and seeding the scaffold with cells for in vivo implantation aiming to replicate the properties of autogenous bone and decrease the need for invasive harvesting Bone marrow contains a heterogenous population of progenitor cells such as Mesenchymal stem cells (MSC),hematopoietic stem cells (HSC) and endothelial progenitor cells in addition to several growth factors, including platelet-derived growth factor (PDGF), transforming growth factor-beta (TGF-b), and bone morphogenetic protein (BMP)-2 and BMP-7, which are known to have anabolic and anti-inflammatory effects. Concentration of the mononuclear cell fraction (MNC) of bone marrow aspirate ( which includes MSCs) by density gradient centrifugation process to remove erythrocytes, granulocytes, platelets and immature myeloid precursors to form Bone Marrow Aspirate Concentrate (BMAC) is considered important step in BTE. .

Many clinical studies proved the use of Bone Marrow Aspirate Concentrate for treatment of osseous defects and cartilage defects due to the ability of MSCs to differentiate into osteoblasts, chondroblasts or adipocytes.

The mesenchymal stem cells (MSCs) are highly biologically competent as they possess the ability to adhere on plastic (scaffolds) in vitro, form colony forming fibroblasts (CFU) and differentiate into mesenchyme lineages ( adipocytes, osteocytes, chondrocytes, tenocytes, myocytes) in addition to their potential of self renewal and promotion of hematopoiesis. Also, they suppress alloresponse after transplantation .

Scaffolds are support structures used in tissue engineering to allow 3D growth of cells in an organized way and can be classified into natural (such as collagen plug) , synthetic aliphatic polyesters such as polycaprolactone (PCL), polyglycolic acid (PGA) and polylactic acid (PLA) and their copolymers and derivatives and composite scaffold which are made by combining bioceramics with polymers or xenogenic biomaterials together with bioceramics or polymers .

ELIGIBILITY:
Inclusion Criteria:

* Patient who require horizontal ridge augmentation in the aesthetic zone (Maxillary anterior and premolar area) with defect size of one or two lost teeth.
* Patients in the age range of 18 years and above.
* ASA physical status I and II.
* Patients willing to be a part of the study and ready to give their consent in writing for the same.

Exclusion Criteria:

* Local criteria:

  * Untreated gingivitis, periodontitis.
  * Insufficient oral hygiene.
  * Previous radiation therapy the head and neck neoplasia, or bone augmentation to implant site.

Systemic criteria:

* Systemic disorders.
* Smoking.
* Bone pathology.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Bone Width gain | 6 months
  The width of the augmented alveolar ridge measured from the Cone Beam Computed Tomography in millimeters

SECONDARY OUTCOMES:
Percentage of bone formation in the bone biopsy | 6 months
  Bone biopsy is obtained after 6 months and subjected to histomorphometric analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo university, Cairo, Egypt

REFERENCES:
- [Background] Chahla J, Dean CS, Moatshe G, Pascual-Garrido C, Serra Cruz R, LaPrade RF. Concentrated Bone Marrow Aspirate for the Treatment of Chondral Injuries and Osteoarthritis of the Knee: A Systematic Review of Outcomes. Orthop J Sports Med. 2016 Jan 13;4(1):2325967115625481. doi: 10.1177/2325967115625481. eCollection 2016 Jan. PMID 26798765
- [Background] Cotter EJ, Wang KC, Yanke AB, Chubinskaya S. Bone Marrow Aspirate Concentrate for Cartilage Defects of the Knee: From Bench to Bedside Evidence. Cartilage. 2018 Apr;9(2):161-170. doi: 10.1177/1947603517741169. Epub 2017 Nov 10. PMID 29126349
- [Background] Dominici M, Le Blanc K, Mueller I, Slaper-Cortenbach I, Marini F, Krause D, Deans R, Keating A, Prockop Dj, Horwitz E. Minimal criteria for defining multipotent mesenchymal stromal cells. The International Society for Cellular Therapy position statement. Cytotherapy. 2006;8(4):315-7. doi: 10.1080/14653240600855905. PMID 16923606
- [Background] Jager M, Jelinek EM, Wess KM, Scharfstadt A, Jacobson M, Kevy SV, Krauspe R. Bone marrow concentrate: a novel strategy for bone defect treatment. Curr Stem Cell Res Ther. 2009 Jan;4(1):34-43. doi: 10.2174/157488809787169039. PMID 19149628
- [Background] McAllister BS, Haghighat K. Bone augmentation techniques. J Periodontol. 2007 Mar;78(3):377-96. doi: 10.1902/jop.2007.060048. PMID 17335361
- [Background] Sanz M, Dahlin C, Apatzidou D, Artzi Z, Bozic D, Calciolari E, De Bruyn H, Dommisch H, Donos N, Eickholz P, Ellingsen JE, Haugen HJ, Herrera D, Lambert F, Layrolle P, Montero E, Mustafa K, Omar O, Schliephake H. Biomaterials and regenerative technologies used in bone regeneration in the craniomaxillofacial region: Consensus report of group 2 of the 15th European Workshop on Periodontology on Bone Regeneration. J Clin Periodontol. 2019 Jun;46 Suppl 21:82-91. doi: 10.1111/jcpe.13123. PMID 31215114
- [Background] Seibert JS. Reconstruction of deformed, partially edentulous ridges, using full thickness onlay grafts. Part I. Technique and wound healing. Compend Contin Educ Dent (Lawrenceville). 1983 Sep-Oct;4(5):437-53. No abstract available. PMID 6578906
- [Background] Seibert JS. Reconstruction of deformed, partially edentulous ridges, using full thickness onlay grafts. Part II. Prosthetic/periodontal interrelationships. Compend Contin Educ Dent (Lawrenceville). 1983 Nov-Dec;4(6):549-62. No abstract available. PMID 6321099
- [Background] Shanbhag S, Suliman S, Pandis N, Stavropoulos A, Sanz M, Mustafa K. Cell therapy for orofacial bone regeneration: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:162-182. doi: 10.1111/jcpe.13049. PMID 30623455